CLINICAL TRIAL: NCT00697216
Title: Study Comparing the Immunogenicity and Reactogenicity of GSK Biologicals' HBV-MPL Vaccine Injected According to a 0, 6 Months Schedule With That of Engerix™-B Injected as a 0, 1, 6 Months Schedule in a Healthy Adult Population (15-40 Years)
Brief Title: Immunogenicity and Safety of GSK Biologicals' HBV-MPL Vaccine and Engerix™-B in Healthy Adults (15-40 Yrs).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/027
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Recombinant hepatitis B vaccine; Adjuvanted hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 2-dose intramuscular injection
  Arms: Group A
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group B

SUMMARY:
This study evaluates the safety and immunogenicity of the candidate HBV-MPL vaccine administered to healthy adults aged from 15 to 40 years, according to a 0, 6- month vaccination schedule, with Engerix™-B as control administered at 0, 1, 6 months.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Age: between 15 and 40 years old.
* Good physical condition as established by clinical examination and history taking at the time of entry.
* Female participants who are at risk to become pregnant will be on a contraceptive programme if necessary during the study period.
* Written informed consent obtained from the subjects aged between 18 and 40 and from the parents/tutor when the subjects are aged between 15 and 17 years.

Exclusion Criteria:

* Positive titres at screening for anti-HBs antibodies.
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Any chronic drug treatment, including any treatment with immunosuppressive drugs, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous participation in any other clinical trial.
* Previous vaccination with a hepatitis B vaccine.
* Previous vaccination with an MPL containing vaccine.
* Administration of immunoglobulins in the past 6 months and during the whole study period
* Simultaneous vaccination one week before and one week after each dose of the study vaccine

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 340 (Actual)
Dates: Start 1997-03; Primary Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | Month 7

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At months 1, 2, 6, 7 and 12
Occurrence, intensity and relationship to vaccination of solicited local and general symptoms | 4-day follow-up period after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | 31-day follow-up after vaccination
Occurrence and relationship to vaccination of Serious Adverse Events (SAEs) | During the study period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Clinical Trials Call Center, Brussels, Belgium
- GSK Clinical Trials Call Center, Copenhagen, Denmark